CLINICAL TRIAL: NCT00087061
Title: Oral ST1481 in Adults With Malignant Glioma: A Phase I-II Clinical Trial
Brief Title: Gimatecan in Treating Patients With Recurrent or Progressive Primary Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: SIGMATAU-ST-01-402; UCLA-0403029-01; SIGMATAU-ST-01-402
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2005-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — ST 1481

INTERVENTIONS:
Drug: gimatecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gimatecan, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gimatecan in treating patients with recurrent or progressive primary malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of gimatecan in patients with recurrent or progressive primary malignant glioma treated with or without concurrent enzyme-inducing anticonvulsant drugs.
* Determine whether this drug has sufficient activity to warrant further development in these patients. (phase II)

Secondary

* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the pharmacokinetic behaviors of this drug in these patients.
* Correlate the principal toxic effects with the pertinent pharmacokinetic parameters of this drug in these patients.
* Determine the antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study. Patients are stratified according to the concurrent use of enzyme-inducing anticonvulsant drugs (yes vs no).

* Phase I: Patients receive oral gimatecan once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gimatecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive gimatecan as in phase I at the MTD. Patients are followed for at least 1 month and then every 2 months thereafter.

PROJECTED ACCRUAL: Approximately 30-83 patients (30-42 for phase I [15-21 per stratum] and 21-41 for phase II) will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma (glioblastoma multiforme, anaplastic astrocytoma, or anaplastic oligodendroglioma)

  * Recurrent or progressive primary CNS neoplasm by contrast-enhanced MRI
* Tumor progression after prior surgery, radiotherapy, or chemotherapy
* Measurable or evaluable disease
* Failed prior standard curative or palliative therapy (phase I only)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGPT and SGOT ≤ 1.5 times upper limit of normal (ULN) (3 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Bilirubin normal

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No myocardial infarction with the past year
* No heart failure (including cardiac insufficiency controlled by digitalis and diuretics)
* No irreversible arrhythmias requiring permanent medication
* No uncontrolled hypertension

Gastrointestinal

* No gastrointestinal dysfunction that would alter absorption or motility, such as any of the following:

  * Active peptic ulcer
  * Inflammatory bowel disease
  * Known intolerance to lactose
  * Malabsorption syndromes
  * Intestinal sub-occlusion

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No active infection
* No mentally incapacitated patients
* No other concurrent severe disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No more than 1 prior chemotherapy regimen
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed if dose stable for the past 2 weeks
* No concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 3 weeks since prior surgical resection
* No prior gastrointestinal surgery that would affect drug absorption

Other

* More than 4 weeks since prior participation in any other investigational drug study
* More than 72 hours since prior systemic antibiotics
* No concurrent H2 antagonists, antacids, or proton pump inhibitors

  * If any of these therapies are necessary, ≥ 3 hours must elapse after gimatecan administration
* No other concurrent anticancer therapy
* No other concurrent investigational drugs
* No other concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F. Cloughesy, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States